CLINICAL TRIAL: NCT01319292
Title: To Investigate the Prevalence of Children Asthma in China and Compare With That of the Last 20 Years
Brief Title: To Investigate the Prevalence of Children Asthma in China
Status: Completed | Type: Observational
Sponsor: Capital Institute of Pediatrics, China (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Chen Yuzhi, Professor, Capital Institute of Pediatrics, China
Other Study IDs: MISP38877
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Asthma children: children with asthma symptoms through screening
- normal children: children without symptoms of asthma

SUMMARY:
Asthma is the most common chronic respiratory disease in children and has much effect on their life and study, which leads to huge economic burden and pressure to the whole families. Some children will develop into adult patients so that asthma can be the life-long vigorous trouble. In recent years, the prevalence rate of children asthma is increasingly going up worldwide. The prevalence rate in last 12 months reported in USA, United Kingdom, Australia, New Zealand was between 12% to 30%.

Center for Asthma Prevention and Education of Capital Institute of Pediatrics investigated the national asthma prevalence in 900 thousands children in 27 provinces and cities, which average rate was 0.11% to 2.03% in 1990. In 2000, we investigated it again in 31 provinces(43 cities) and the average national children asthma prevalence rate was 1.97%(0.25% to 4.63%) which was much higher than that in 1990.

DETAILED DESCRIPTION:
1. Objectives

   1. To investigate the national children(0-14 years old)asthma prevalence;
   2. To compare the prevalence rate between that in 1990 and 2000;
   3. To analyse the asthma manifestations including the ages, seasons, causes, trigger and hereditary factors and their impact on the asthma patients, families and society;
   4. To identify the risk factors by questionnaires in case-control research.
2. Study Design / Clinical Plan

   1. The screening stage: to distinguish suspected asthma from the children age from 0 to 14 years old.
   2. To obtain identified asthma from the suspected asthma.
   3. To evaluate the prevalence and severe degree of 0 to 14-year-old children asthma and gain the main risk factors by case-control research.

ELIGIBILITY:
Inclusion Criteria:

* children age from 0 to 14 years

Exclusion Criteria:

* none

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children age from 0 to 14 years in big cities in China
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
prevalence of asthma | Apr 2013

SECONDARY OUTCOMES:
prevalence of allergic rhinitis | Apr 2013

CONTACTS AND LOCATIONS:
Overall Officials: YuZhi Chen, professor, Study Chair — Capital Institute of Pediatrics, China